CLINICAL TRIAL: NCT05421715
Title: Preliminary Study for the Evaluation of Teleduc-diab Additional Remote Digitalcare Effects in Adolescents With Poorly Controled Type 1 Diabetes
Brief Title: Remote Digital Care Effects in Adolescents With Type 1 Diabetes
Acronym: TELEDUC-DIAB1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0617
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: type1diabetes
Keywords: glucose control; patient therapeutic education; mobile application; remote digital care; adolescents; teenagers

STUDY DESIGN:
Intervention Model Description: Monocentric longitudinal prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALL ADOLESCENTS (Experimental): For all adolescents, the proposed treatment consists, in addition to conventional care,an individual digital care and education(TELEDUC-DIAB)for 6 months using digital devices (myDiabby + Kidia).
  Interventions: Other: TELEDUC-DIAB

INTERVENTIONS:
Other: TELEDUC-DIAB — * Systematic monthly remote monitoring between traditional face-to-face consultations by a medical researcher using Kidia and My Diabby digital devices:
    * With downloading by the adolescent of all data on My Diabby platform (clinical data from diabetes monitoring)
    * Evaluation of adverse events related to the treatment of diabetes (hospitalizations and concomitant treatment)
    * Analysis of data collected via My Diabby and Kidia: glycemic balance, captured data, connection frequency, alerts and alarms, diabetes knowledge)
    * The proposal of a therapeutic education session according to the needs of the adolescent via the Kidia application
    * Treatment adaptation
  * A follow-up in case there is an alert identified by the teenager, the relative or My Diabby/caregiver
    * The medical orientation of the patient according to the needs identified
    * A proposal for a therapeutic education session according to the needs of the adolescent via the Kidia application

SUMMARY:
Pilot study to evaluate effects of an experimental additional remote digital care (TELEDUC-DIAB) to adolescents with poorly controlled type 1 diabetes using digital monitoring platform and educative app

DETAILED DESCRIPTION:
The use of digital technologies for the support and monitoring of diabetes have gradually become essential in recent years. The scientific literature reveals contrasting effects of digital and mobile technologies, both on adolescents with T1D (type 1 diabetes) and on their relatives. While the majority of studies have focused on connected devices for continuous blood glucose measurement, the specific effects of other tools, such as those of mobile patient therapeutic education applications or medical telemonitoring, are to this day still poorly documented or even unknown.

The study aim to describe the evolution of the glycemic control of adolescents with poorly controled type 1 diabetes during6 months individual TELEDUC-DIAB remote digital care in addition to their conventional follow-up.

The Medical-educational care (TELEDUC-DIAB) consist of:

* a personalized intensified remote care with a healthcare professional
* myDiabby platform: remote monitoring device integrating a data collection platform and systematized monitoring by alarms
* the Kidia application = a patient therapeutic education mobile application: developed by the Enfance, Adolescence et Diabète association, is a mobile application that patients can personalize (avatar,...) and help them understand and empower to deal with their diabetes.

This project offers original and innovative complementary monitoring: remotely, adapted to the specific needs of adolescents and aimed at improving glycemic control by developing self-efficacy and autonomy in adolescents in the management of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent aged ≥12 and <18, with primary type 1 diabetes detected for at least 12 months, treated with multi-injection insulin or insulin pump
* Glycated hemoglobin greater than or equal to 8% for more than 3 months
* Use a continuous interstitial glucose recording system (CGM)
* Have at least one parent/guardian with a significant caregiver role in the management of the adolescent's diabetes (as determined by the investigator) participating in the study
* Have digital media compatible with the digital applications of the TELEDUC- DIAB (Mobile phone and computer)

Exclusion Criteria:

• Other pathologies associated with diabetes which, according to the investigator, could interfere with glycemic control or the management of adolescent diabetes (examples: secondary diabetes, cystic fibrosis, Down syndrome; transplants, corticosteroid therapy, etc.)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of glycemic control hemoglobin (HbA1c) between inclusion and 6 months | 6 months after inclusion
  Glycated hemoglobin (HbA1c) is currently the universally recognized biological marker for monitoring diabetes.
  Glycated hemoglobin levels will be measured at inclusion, then 6 months after inclusion : a ratio will be deduced 6 months after inclusion with those two measures.

SECONDARY OUTCOMES:
Evolution of adherence to TELEDUC-DIAB management between inclusion and 6 months | 6 months after inclusion
  Non-adherence to the program will be determined if:
  * <80% of interstitial blood glucose is entered by the adolescent on the app over the last 14 days
  * For adolescents with an insulin pump: average duration between 2 catheter changes greater than 3 days
  * Monthly frequency of use of the TELEDUC-DIAB device :
    * < 4 monthly connections to the download platform
    * <1 monthly connection to the KIDIA application
    * <1 monthly telemonitoring connection with the professional
Evolution of knowledge about diabetes and glycemic targets between inclusion and T6 months | 6 months after inclusion
  an open question is asked to the participant each months of the study: "describe what glycated hemoglobin (hb1AC) is and the ideal ranges in which capillary blood glucose and hemoglobin measurements glycated must be located" Correctly answering these 3 key questions is associated with better glycemic control.
  Each question will be scored by 0 (wrong answer or no answer), 0.5 (incomplete answer) and 1 (correct and complete answer).

CONTACTS AND LOCATIONS:
Overall Officials: Maeva TALVARD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital TOULOUSE, Toulouse, France